CLINICAL TRIAL: NCT03198741
Title: COmparison of Mono- Versus Dual antiPlatelet Therapy During 6-12 Months After New Generation Drug Eluting Stent Implantation for Prevention of Gastrointestinal Injury Evaluated by Ankon Magnetically Controlled Capsule Endoscopy
Brief Title: Mono- Versus Dual antiPlatelet Therapy During 6-12 Months After New Generation Drug Eluting Stent Implantation
Acronym: OPT-PEACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Collaborators: Changhai Hospital (Other); ANKON medical technologies (Shanghai)Co.,LTD (Unknown)
Responsible Party: Principal Investigator, Han Yaling, Director of the Cardiology department, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYNH-20170602
Record Dates: First submitted 2017-06-19; First posted 2017-06-26 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Gastrointestinal Injury; Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aspirin+clopidogrel (Active Comparator): Open label clopidogrel (75mg/d) plus aspirin (100mg/d) for first 6 months after enrollment. At 6 months (±2 weeks),continue aspirin + clopidogrel (12-month DAPT group).The treatments between 6 and 12 months are double-blinded.
  Evaluation of gastric and intestinal mucosal lesions by AMCE will be performed at the time of screening, randomization (at 6 months ±2 weeks) and 6 months thereafter (at 12 months ±2 weeks).
  Interventions: Drug: Aspirin + clopidogrel
- Aspirin (Experimental): Open label clopidogrel (75mg/d) plus aspirin (100mg/d) for first 6 months after enrollment. At 6 months (±2 weeks),receive aspirin + placebo (aspirin monotherapy group) for an additional 6 months. The above treatments between 6 and 12 months are double-blinded.
  Evaluation of gastric and intestinal mucosal lesions by AMCE will be performed at the time of screening, randomization (at 6 months ±2 weeks) and 6 months thereafter (at 12 months ±2 weeks).
  Interventions: Drug: Aspirin monotherapy
- Clopidogrel (Experimental): Open label clopidogrel (75mg/d) plus aspirin (100mg/d) for first 6 months after enrollment. At 6 months (±2 weeks),receive clopidogrel + placebo (clopidogrel monotherapy group) for an additional 6 months. The above treatments between 6 and 12 months are double-blinded.
  Evaluation of gastric and intestinal mucosal lesions by AMCE will be performed at the time of screening, randomization (at 6 months ±2 weeks) and 6 months thereafter (at 12 months ±2 weeks).
  Interventions: Drug: Clopidogrel monotherapy

INTERVENTIONS:
Drug: Aspirin + clopidogrel — After randomization(6 months±2 weeks after enrollment),receive aspirin 100mg/d + clopidogrel 75mg/d for an additional 6 months. The above treatments between 6 and 12 months are double-blinded.
  Arms: Aspirin+clopidogrel
Drug: Clopidogrel monotherapy — After randomization(6 months±2 weeks after enrollment),receive clopidogrel 75mg/d + placebo (clopidogrel monotherapy group) for an additional 6 months. The above treatments between 6 and 12 months are double-blinded.
  Other Names: Clopidogrel + placebo
  Arms: Clopidogrel
Drug: Aspirin monotherapy — After randomization(6 months±2 weeks after enrollment),receive aspirin 100mg/d + placebo (aspirin monotherapy group) for an additional 6 months. The above treatments between 6 and 12 months are double-blinded.
  Other Names: Aspirin + clopidogrel
  Arms: Aspirin

SUMMARY:
Long-term DAPT is recommended after percutaneous coronary intervention (PCI) in patients with coronary artery disease. However, antiplatelet therapy may have adverse consequences, the most common of which is gastrointestinal mucosal injury with ulceration and bleeding. The extent to which an an abbreviated DAPT strategy reduces gastrointestinal mucosal injury has not been studied, principally due to the lack of sensitive, noninvasive measurements capable of detecting gastrointestinal injury.ANKON® magnetically controlled capsule endoscopy (AMCE) is a non-invasive, active controlled system which affords assessment of the stomach and entire small intestine.The current randomized study will assess gastrointestinal mucosal injury and bleeding via AMCE in patients on three different antiplatelet regimens and establish a gastrointestinal mucosal injury scoring system which may prove useful in guiding optimal antiplatelet agent usage after PCI.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and a platelet P2Y12 receptor inhibitor has become the cornerstone for secondary prevention of coronary artery disease. Long-term DAPT is recommended after percutaneous coronary intervention (PCI) in patients with coronary artery disease to prevent future thrombotic events arising from the stent or untreated coronary lesions. However, antiplatelet therapy may have adverse consequences, the most common of which is gastrointestinal mucosal injury with ulceration and bleeding. The frequency of gastrointestinal complications increases with the duration of DAPT. Studies in patients treated with current generation drug-eluting stents have demonstrated that shortened DAPT regimens reduce the risk of bleeding events with small ischemic risk. However, the optimal duration of DAPT is still controversial. The extent to which an an abbreviated DAPT strategy reduces gastrointestinal mucosal injury has not been studied, principally due to the lack of sensitive, noninvasive measurements capable of detecting gastrointestinal injury.

Endoscopic examination of the gastric mucosa (gastroscopy) has high sensitivity and accuracy to detect gastrointestinal injury and bleeding. However, endoscopy is invasive and thus has no role in screening for sub-clinical gastrointestinal bleeding in patients undergoing PCI. Rather, endoscopy examinations are reserved for patients with active bleeding to identify the location of origin and etiology of the bleed. Moreover, gastroenterologists often refuse to perform gastroscopy in patients on DAPT given the risk of iatrogenic trauma with excessive hemorrhage. To minimize this risk, one or both antiplatelet agents often have to be discontinued for several days prior to the procedure, delaying the diagnosis while increasing the risk of stent thrombosis. Finally, upper endoscopy can only detect pathology related to the stomach and duodenum, as it does not visualize the remainder of the small intestine.

ANKON® magnetically controlled capsule endoscopy (AMCE) is a non-invasive, active controlled system which affords assessment of the stomach and entire small intestine. In the AMCE procedure, the patient swallows a capsule containing an endoscope which is actively maneuvered via magnetic control in the stomach, and then passes through the gastrointestinal track until its ultimate excretion. AMCE has several advantages compared to standard endoscopy. AMCE is noninvasive, painless and convenient, and can be re-administered as necessary. Patient acceptance of AMCE is likely to be substantially higher than standard endoscopy as the procedure involves only swallowing a capsule endoscope, without anesthesia or recovery time. Compared to standard endoscopy, AMCE provides more comprehensive detection of gastrointestinal pathology as it visualizes not only the stomach and duodenum, but the entire small intestine. Finally, discontinuation of antiplatelet drugs during AMCE is not necessary. Because of these advantages, AMCE can be used for screening of gastrointestinal mucosal lesions prior to clinical bleeding, including early detection of small areas of focal and concealed bleeding. Detection of preclinical gastric ulcerations or bleeding may be useful in directing preventative measures, whether gastro-protective therapies or DAPT discontinuation. A large-scale, randomized trial has confirmed that the sensitivity and specificity of AMCE for the detection of focal lesions of the gastrointestinal tract is similar to standard endoscopy. However, the potential utility of AMCE in patients receiving antiplatelet therapy after PCI has not been reported.

The current randomized study will evaluate AMCE as a tool to assess gastrointestinal mucosal injury and bleeding in patients on DAPT; evaluate the relative rates of gastrointestinal injury in patients on three different antiplatelet regimens; and establish a gastrointestinal mucosal injury scoring system which may prove useful in guiding optimal antiplatelet agent usage after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with age of 18-80 years;
2. Presentation with silent ischemia, stable angina, or non-ST-segment elevation acute coronary syndrome with GRACE score <140 on admission;
3. PCI only with implantation of current generation drug-eluting stent(s) for coronary artery disease during the present admission [current generation DES refers to DES with thin cobalt-chromium or platinum-chromium struts, with a durable or biodegradable polymer eluting a rapamycin-analogue antiproliferative agent. The current major DES available in China market include: EXCEL and EXCEL 2 (JW Medical System, Weihai, China), Tivoli（Essen Technology, Beijing, China), Endeavor Resolute (Medtronic Inc., Minnesota, USA), FireHawk (MicroPort Medical (Group) Co., Ltd, Shanghai, China), BuMA (SinoMedical,China),Xience V (Abbott Laboratories, Abbott Park, Illinois, USA), Xience Prime (Abbott Laboratories, Abbott Park, Illinois, USA), Promus Element and Synergy (BostonTechnologies, Massachusetts, USA)].
4. PCI resulted in complete revascularization (successful PCI treatment of all epicardial coronary lesions with diameter stenosis >70% or intermediate lesions with FFR ≤0.80);
5. Intended treatment with dual antiplatelet therapy (aspirin + clopidogrel) after the DES procedure for at least 6 months;
6. Agreement to comply with all study procedures.
7. Written informed consent provided.

Exclusion Criteria:

1. Presentation with STEMI;
2. Left main disease (diameter stenosis >30% );
3. Any prior coronary stent implantation during the last year prior to the index procedure;
4. Implantation of of first-generation drug-eluting stents or bioabsorbable scaffolds during the index procedure;
5. Implantation of >4 stents during the index procedure;
6. Any prior stent thrombosis;
7. Any active gastrointestinal bleeding or ulcers, or prior gastrointestinal bleeding or ulcers within the last 24 months;
8. Prior gastrointestinal tract or abdominal surgery other than simple procedures which would not change the gastrointestinal tract anatomy, such as polyp removal, cholecystectomy or appendectomy;
9. Contraindications to the AMCE test, including suspected or known gastrointestinal obstruction, stenosis, fistula, diverticula, etc.; presence of gastrointestinal obstruction symptoms such as pain or dysphagia; inoperative conditions or refusal to undergo abdominal surgery if required (i.e, if the capsule will not pass and cannot be removed by endoscopy)
10. Severe hemorrhoids (phase 3-4 according to guidelines of American Society of Colon and Rectal Surgery);
11. LVEF <0.40 on admission according to cardiac ultrasound;
12. Renal dysfunction (eGFR <30ml/min/1.73m2);
13. Active hepatitis or ALT >3 times upper limits of normal on admission;
14. Uncontrolled severe hypertension (>180/110mmHg);
15. Hemoglobin <100 g/L;
16. Platelet count <100×109/L;
17. Planned use of a proton pump inhibitor, gastric mucosa protectant or any other antacid agent after study enrollment；
18. Required use of oral anticoagulation (warfarin or other factor II or factor X inhibitors);
19. Inability to take 12-month DAPT for any reason;
20. Mandatory use of >6 month DAPT (i.e. contraindication to aspirin or clopidogrel monotherapy after 6 months);
21. Any comorbidity with estimated survival time <12 months (e.g. progressive cancer, chronic obstructive lung disease, etc.);
22. Any contraindication to MRI examination, including implantation of an MRI-incompatible pacemaker, defibrillator, or other ferromagnetic material; etc.
23. Pregnant or plan to be pregnant within 1 year;
24. Any condition that may interfere with any study procedures, such as dementia, immobility, alcohol use, etc.;
25. Planned surgery within 1 year;
26. Taking iron supplement;
27. Participating in any other clinical trial of an investigational drug or device that has not met its primary endpoint.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 783 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal mucosal Injury (erosion, ulceration or bleeding) | 12 months after enrollment (i.e. 6 months after randomization)
  Detected by AMCE

SECONDARY OUTCOMES:
The severity of gastric and intestinal mucosal lesions | During the first 6 months after study enrollment (prior to randomization)
  Detected by AMCE and calculated with a score system
The severity of gastric and intestinal mucosal lesions | After randomization (i.e. between 6 months and 12 months after study enrollment)
  Detected by AMCE and calculated with a score system
Clinical indicated bleeding of the upper gastrointestinal tract | During 6 months after study enrollment (prior to randomization)
  1. Hematemesis is defined as vomiting of blood or blood clots, and generally indicates bleeding of the upper gastrointestinal tract.
  2. Hematochezia is the passage of fresh blood per anus, usually in or with stools, and typically signifies lower GI tract bleeding.
  3. Melena is the passage of black, tarry stool and typically signifies upper tract GI bleeding.
  4. The positive fecal occult blood refers to blood in the feces that is not visibly apparent (unlike other types of blood in stool such as melena or hematochezia).
Clinical indicated evident gastrointestinal hemorrhage | After randomization (i.e. between 6 months and 12 months after study enrollment)
  1. Hematemesis is defined as vomiting of blood or blood clots, and generally indicates bleeding of the upper gastrointestinal tract.
  2. Hematochezia is the passage of fresh blood per anus, usually in or with stools, and typically signifies lower GI tract bleeding.
  3. Melena is the passage of black, tarry stool and typically signifies upper tract GI bleeding.
  4. The positive fecal occult blood refers to blood in the feces that is not visibly apparent (unlike other types of blood in stool such as melena or hematochezia).
Clinical indicated gastrointestinal hemorrhage | 12 months after enrollment (i.e. 6 months after randomization)
  1. Hematemesis is defined as vomiting of blood or blood clots, and generally indicates bleeding of the upper gastrointestinal tract.
  2. Hematochezia is the passage of fresh blood per anus, usually in or with stools, and typically signifies lower GI tract bleeding.
  3. Melena is the passage of black, tarry stool and typically signifies upper tract GI bleeding.
  4. The positive fecal occult blood refers to blood in the feces that is not visibly apparent (unlike other types of blood in stool such as melena or hematochezia).
Gastrointestinal symptoms | 12 months after enrollment (i.e. 6 months after randomization)
  pain, nausea/vomiting, dysphagia, other discomfort
All bleeding | 12 months after enrollment (i.e. 6 months after randomization)
  BARC types 1-5
Target lesion failure | 12 months after enrollment (i.e. 6 months after randomization)
  TLF: cardiac death, target-vessel MI, or clinically-driven target lesion revascularization
Net adverse clinical events | 12 months after enrollment (i.e. 6 months after randomization)
  NACE, defined as TLF or BARC type 2-5 bleeding
Stent thrombosis | 12 months after enrollment (i.e. 6 months after randomization)
  ARC definite, probable, or definite/probable

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, PhD, Principal Investigator — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Wang X, Bao D, Liao Z, Li J, Han X, Wang H, Xu K, Li Z, Stone GW, Han Y. Optimal antiplatelet therapy for prevention of gastrointestinal injury evaluated by ANKON magnetically controlled capsule endoscopy: Rationale and design of the OPT-PEACE trial. Am Heart J. 2020 Oct;228:8-16. doi: 10.1016/j.ahj.2020.06.004. Epub 2020 Jun 15. PMID 32745734
- [Background] Han Y, Liao Z, Li Y, Zhao X, Ma S, Bao D, Qiu M, Deng J, Wang J, Qu P, Jiang C, Jia S, Yang S, Ru L, Feng J, Gao W, Huang Y, Tao L, Han Y, Yang K, Wang X, Zhang W, Wang B, Li Y, Yang Y, Li J, Sheng J, Ma Y, Cui M, Ma S, Wang X, Li Z, Stone GW. Magnetically Controlled Capsule Endoscopy for Assessment of Antiplatelet Therapy-Induced Gastrointestinal Injury. J Am Coll Cardiol. 2022 Jan 18;79(2):116-128. doi: 10.1016/j.jacc.2021.10.028. Epub 2021 Nov 6. PMID 34752902
- [Derived] He C, Li Y, Jiang X, Jiang MN, Zhao XX, Ma SR, Bao D, Qiu MH, Deng J, Wang JH, Qu P, Jiang CM, Jia SB, Yang SQ, Ru LS, Feng J, Gao W, Huang YH, Tao L, Han Y, Yang K, Wang XY, Zhang WJ, Wang BM, Li Y, Yang YL, Li JX, Sheng JQ, Ma YT, Cui M, Ma SC, Wang XZ, Li ZS, Liao Z, Han YL, Stone GW. Progression of Gastrointestinal Injury During Antiplatelet Therapy After Percutaneous Coronary Intervention: A Secondary Analysis of the OPT-PEACE Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2343219. doi: 10.1001/jamanetworkopen.2023.43219. PMID 37976067